CLINICAL TRIAL: NCT05420181
Title: The Effect of Prolonged Overnight Fast on Postprandial Energy Metabolism and Skeletal Muscle Anabolic Sensitivity in Healthy Humans
Brief Title: Prolonged Overnight Fast, Energy Metabolism and Skeletal Muscle Anabolic Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Kostas Tsintzas, Professor of Human Physiology, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 289-1904
Record Dates: First submitted 2022-04-08; First posted 2022-06-15 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Time Restricted Feeding
Keywords: Energy metabolism; skeletal muscle; protein synthesis
MeSH Terms: conditions — Intermittent Fasting

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short Fast (Other): Participants will fast overnight for a period of 10 hours
  Interventions: Other: Short 10hr fast
- Long fast (Other): Participants will fast overnight for a period of 16 hours
  Interventions: Other: Long 16h fast

INTERVENTIONS:
Other: Short 10hr fast — Participants will fast from 11pm the night before the study day
  Arms: Short Fast
Other: Long 16h fast — Participants will fast from 5pm the night before the study day
  Arms: Long fast

SUMMARY:
Recent research shows that timing of nutritional intake and daily periods of fasting may have important health effects. In humans, limiting daily food intake to a narrow window (typically ~8 hours) can bring about some beneficial changes in blood concentrations of fats, sugar and the hormone insulin. It is thought that many of these changes are due to the prolonged daily fasting periods and humans will have regularly experienced prolonged fasting periods throughout evolution. In the modern era, food access is widely available and it is not uncommon for the time between breakfast and a late night snack to exceed 14 hours. We have recently shown that extending habitual daily periods of fasting to 16 hours per day also improves the ability of skeletal muscle to take up amino acids, the building blocks of protein. We are interested in studying whether a single episode of prolonged overnight fast (~16 hours), when compared to a normal overnight fast of 10 hours, is sufficient to stimulate skeletal muscle protein synthesis in response to dietary protein ingestion in healthy humans.

DETAILED DESCRIPTION:
There is a growing interest in the cardiometabolic benefits of various intermittent fasting paradigms (such as alternate day fasting and the 5:2 fast diet), where periods of normal energy intake are punctuated by periods of energy restriction or fasting. A recent alternative to these protocols is time-restricted feeding (TRF), which limits daily food/energy intake to a narrow window (typically 8 to 10h). The major strength of TRF is that it extends the duration of overnight fast without limiting normal calorie intake. Recent evidence from both animal and human studies have shown that habitual daily periods of fasting of as little as 16h can reduce fasting insulin and triglycerides levels, protect against excessive body weight gain in response to high fat and sucrose diets, better maintain fat-free mass, and improve beta-cell responsiveness. We recently completed a 2-week TRF intervention study using the 8h fed (between 8am and 4pm)/16h fast protocol in healthy individuals and found improvements in insulin sensitivity and skeletal muscle uptake of branched chain amino acids. As we did not make measurements of muscle protein synthesis, it is not known whether a single episode of prolonged overnight fast (~16h) is sufficient to elicit improvements in insulin sensitivity and stimulate skeletal muscle protein synthesis in response to dietary protein ingestion. The aim of the proposed study is to investigate the effect of prolonged overnight fast (16h vs. 10h) on postprandial energy metabolism and skeletal muscle protein synthesis in healthy humans.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-35yrs
* healthy
* non-smoking
* physically active
* no excessive weight loss in past 6 months
* body mass index between 18 and 27 kg.m-2

Exclusion Criteria:

* body mass index under 18 and over 27 kg.m-2
* sedentary
* screening bloods out of range
* excessive weight loss in the past 6 months
* irregular eating patterns

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Whole body Insulin sensitivity | 3 hours
  Postprandial blood glucose and serum insulin concentrations will be used to compute the Matsuda index of whole body insulin sensitivity. Postprandial blood glucose and serum insulin concentrations will be measured every 15mins for 3 hours in response to ingestion of a protein and dextrose drink. Serum insulin concentration (mIU/l) will be measured either with an enzyme linked immunosorbent assay or a radioimmuno assay. Blood glucose will be measured using the glucose oxidase method.
Glycemic responses | 3 hours
  Postprandial blood glucose incremental area under the curve( iAUC)
Insulinaemic responses | 3 hours
  Postprandial blood insulin iAUC
Index of skeletal muscle protein synthesis (A) | 3 hours
  Skeletal muscle branched chain amino acid uptake using postprandial arteriovenous differences.
Index of skeletal muscle protein synthesis (B) | 3 hours
  Muscle protein synthesis will be measured 3 hours after ingestion of a protein and dextrose drink in which the milk protein has been intrinsically labelled with [1-13C]phenylalanine. The investigators will measure [13C]phenylalanine incorporation into the muscle myofibrillar protein pool during the 3 hour period from a muscle biopsy sample taken pre ingestion of the drink and a muscle biopsy taken 3 hours post ingestion. This will give a rate (%/hour) of muscle protein synthesis.

SECONDARY OUTCOMES:
Skeletal muscle insulin sensitivity | 3 hours
  Postprandial arteriovenous differences in glucose concentration. Blood glucose in arterialised and deep venous blood across the forearm will be measured using the glucose oxidase method.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hatori M, Vollmers C, Zarrinpar A, DiTacchio L, Bushong EA, Gill S, Leblanc M, Chaix A, Joens M, Fitzpatrick JA, Ellisman MH, Panda S. Time-restricted feeding without reducing caloric intake prevents metabolic diseases in mice fed a high-fat diet. Cell Metab. 2012 Jun 6;15(6):848-60. doi: 10.1016/j.cmet.2012.04.019. Epub 2012 May 17. PMID 22608008
- [Background] Chaix A, Zarrinpar A, Miu P, Panda S. Time-restricted feeding is a preventative and therapeutic intervention against diverse nutritional challenges. Cell Metab. 2014 Dec 2;20(6):991-1005. doi: 10.1016/j.cmet.2014.11.001. PMID 25470547
- [Background] Moro T, Tinsley G, Bianco A, Marcolin G, Pacelli QF, Battaglia G, Palma A, Gentil P, Neri M, Paoli A. Effects of eight weeks of time-restricted feeding (16/8) on basal metabolism, maximal strength, body composition, inflammation, and cardiovascular risk factors in resistance-trained males. J Transl Med. 2016 Oct 13;14(1):290. doi: 10.1186/s12967-016-1044-0. PMID 27737674
- [Background] Sutton EF, Beyl R, Early KS, Cefalu WT, Ravussin E, Peterson CM. Early Time-Restricted Feeding Improves Insulin Sensitivity, Blood Pressure, and Oxidative Stress Even without Weight Loss in Men with Prediabetes. Cell Metab. 2018 Jun 5;27(6):1212-1221.e3. doi: 10.1016/j.cmet.2018.04.010. Epub 2018 May 10. PMID 29754952
- [Background] Jones R, Pabla P, Mallinson J, Nixon A, Taylor T, Bennett A, Tsintzas K. Two weeks of early time-restricted feeding (eTRF) improves skeletal muscle insulin and anabolic sensitivity in healthy men. Am J Clin Nutr. 2020 Oct 1;112(4):1015-1028. doi: 10.1093/ajcn/nqaa192. PMID 32729615